CLINICAL TRIAL: NCT05580354
Title: A Prospective, Single Center Clinical Study to Examine the Safety and Efficacy of BCG Combined With Tislelizumab as Treatment for BCG-untreated Patients With High-grade Non-muscle-invasive Bladder Cancer
Brief Title: Safety and Efficacy of BCG Combined With Tislelizumab for BCG-untreated Patients With High-risk Non-muscle Invasive Bladder Cancer
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPARE-007
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Non-muscle-invasive Bladder Cancer
Keywords: Non-muscle-invasive Bladder Cancer; Tislelizumab; BCG
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms | interventions — tislelizumab

STUDY DESIGN:
Intervention Model Description: BCG combined with Tislelizumab
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): Patients will receive 17 cycles of Tislelizumab (200mg per cycle) in combination with BCG (6-week induction course of 120mg followed by maintenance with 3 weekly infusions of 120mg at months 3,6,12).
  Interventions: Drug: BCG combined with Tislelizumab

INTERVENTIONS:
Drug: BCG combined with Tislelizumab — Patients will receive 17 cycles of Tislelizumab (200mg per cycle) in combination with BCG (6-week induction course of 120mg followed by maintenance with 3 weekly infusions of 120mg at months 3,6,12).

SUMMARY:
For patients with high-risk non-muscle-invasive bladder cancer (NMIBC), intravesical therapy of BCG is the standard treatment proved to reduce the risk of recurrence and progression. However, there are patients failed to complete the whole treatment due to the long period and some patients showed no response to BCG or suffered tumor progression after BCG treatment. The aim of this study is to examine the efficacy and safety of intravesical therapy of BCG combined with PD-1 monoclonal antibody as the treatment of high-risk NMIBC patients without BCG treatment. At the same time, transcriptome sequencing is used to analyze the correlation between the efficacy of the treatment and the level of immune cell infiltration and tumor molecular subtypes.

DETAILED DESCRIPTION:
Bladder cancer is a common malignant tumor, with non-muscle-invasive bladder cancer (NMIBC) accounting for approximately 75% of bladder cancer patients. Of these NMIBC patients, 50-70% have tumor recurrence and 15% have tumor progression, thus most patients may require prolonged cystoscopy and therapeutic intervention. According to the EAU guideline, intravesical therapy of BCG is the standard treatment of high-risk NMIBC patients, as it reduces the risk of tumor recurrence and progression. There has long been controversial about the dosage and period of BCG treatment and long-term BCG treatment may cause frequent adverse effects such as hematuria and urinary frequency，because of which many patients failed to complete the whole period of treatment. Also, some patients showed no response to BCG and underwent tumor progression after BCG treatment. Based on the above considerations, trying to improve the treatment for NMBIC patients is important. Recent study showed that the rate of BCG response and tumor recurrence after BCG treatment may be related to PD-L1 expression, indicating that the therapeutic effect of BCG treatment combined with ICIs remains to be explored. Besides, since the molecular subtype of NMIBC has not been well standardized, and molecular subtype may guide treatment options, the correlation between NMIBC molecular subtypes and immunotherapy still remains to be verified by further studies. Since circulating tumour DNA (ctDNA) holding promise as a biomarker for molecular residual disease and relapse, next generation sequencing (NGS) of ctDNA may also benefit treatment options. This trial investigates the safety and efficacy of intravesical therapy of BCG combined with Tislelizumab for BCG-untreated patients with high-risk NMIBC as well as the relationship between the efficacy and tumor subtypes.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤75 years old on day of signing informed consent
* Signing informed consent
* Patients with histologically confirmed high-risk NMIBC after TURBT (Patients with mixed histology, predominantly transitional cells, could be enrolled.) High grade pathology (any of the following conditions)

  * CIS
  * T1
  * >3cm
  * Multifocal
* Patients must be willing to provide a blood sample and a TURBT specimen must be taken at baseline.
* For patients with T1 or suspected incomplete tumor resection after first TURBT, incomplete initial resection or no muscle in original specimen, they should undergo TURBT again within 2-6 weeks.
* No distant metastasis confirmed by CT or MRI in the chest, abdomen, or pelvic cavity within 42 days before treatment.
* ECOG performance status of ≤2
* Life expectancy ≥12 weeks
* Well-controlled blood pressure and within 7 days before treatment <160/95mmHg
* Normal organ function within 7 days before treatment

  * HB≥90 g/L
  * ANC≥1.5×109 /L
  * PLT≥100×109 /L
  * T-BIL≤1.5×ULN
  * ALT, AST≤2.5×ULN
  * eGFR≥ 20ml/min
  * INR, APTT≤1.5× ULN.

Exclusion Criteria:

* Received prior therapies targeting PD-1 or PD-L1.
* Received prior intravesical therapy of BCG.
* Receive any approved anticancer therapy, including systemic and intravesical chemotherapy within 21 days before enrollment.
* Receive any other trial drug or participate in another therapeutic clinical study within 28 days before enrollment.
* History of severe hypersensitivity reactions to other monoclonal antibodies.
* History of other malignancy.
* Active tuberculosis.
* Severe infections occur within 4 weeks prior to enrollment, including but not limited to infectious complications leading to hospitalization, bacteremia, or severe pneumonia.
* A known history of HIV infection.
* Untreated chronic hepatitis B patients or hepatitis B virus carriers whose HBV DNA≥500 IU/mL
* Patients with active hepatitis C
* Participants with active autoimmune diseases or history of autoimmune diseases that may relapse
* Clinically significant cardiovascular disease, including heart disease (NYHA ≥Ⅲ), myocardial infarction, unstable arrhythmia or unstable angina within 3 months before enrollment.
* A known history of LVEF<40%
* Prior allogeneic stem cell transplantation or organ transplantation
* History of interstitial lung disease, noninfectious pneumonitis, or uncontrolled diseases.
* Underlying diseases that the investigator believes are not conducive to study treatment or difficult to explain by drug toxicity or adverse events.
* Receive hormone therapy or other immunosuppressive therapy within 14 days before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2022-10-09 (Estimated); Primary Completion 2024-10-09 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Relapse-Free Survival （RFS） | 12 month
  Relapse-Free Survival （RFS） is defined as the time from enrollment to any event of recurrence or death.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 month
  Overall survival (OS) is defined as the time from enrollment to death from any cause.
Cystectomy-free survival | 12 month
  Cystectomy-free survival is defined as the time from enrollment to radical cystectomy.
Duration of Response (DOR) | 12 month
  Duration of Response (DOR) is defined as the time from CR to any event of recurrence, progression, or death of high-risk NMIBC.
Progression free survival to muscle-invasive or metastatic disease or death. | 12 month
  Progression free survival to muscle-invasive or metastatic disease or death is defined as the time from CR to any event of tumor myometrium invasion, metastasis, or death.
Correlation between biological markers and tumor molecular subtypes and efficacy. | 12 month
  Correlation between biological markers and tumor molecular subtypes and efficacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No